CLINICAL TRIAL: NCT06113081
Title: Real World Experience With Mogamulizumab in the Treatment of Cutaneous T-cell Lymphoma: a Multicenter Observational Study
Brief Title: Real World Experience With Mogamulizumab in the Treatment of Cutaneous T-cell Lymphoma
Acronym: FIL_MOGA
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_MOGA
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous T Cell Lymphoma; Cutaneous T-Cell Lymphoma/Mycosis Fungoides; Cutaneous T-Cell Lymphoma/Sezary Syndrome
Keywords: Cutaneous T Cell Lymphoma; Mycosis Fungoides; Sezary Syndrome; Mogamulizumab; MAVORIC; Retrospective; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patients affected by relapsed/refractory Cutaneous T cell Lymphoma who have received Mogamulizumab in real life setting

SUMMARY:
This study is designed to describe the clinical activity and safety profile of mogamulizumab at standard dose in the treatment of CTCL patients in real world setting

DETAILED DESCRIPTION:
Mogamulizumab (anti-CCR4) has been recently approved and reimbursed in Italy for the treatment of Cutaneous T-cell lymphoma (CTCL) after 1 previous systemic treatment based on the favourable results of the MAVORIC clinical trial. To date, no real-world data on significant series of patients treated routinely with mogamulizumab in clinical practice are available. As real-life data are essential to confirm the preliminary evidence displayed in phase III trials, this study aims at describing the clinical activity and safety profile of mogamulizumab at standard dose in the treatment of CTCL patients in real world settings.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CTCL according to the EORTC 2017 update criteria (Trautinger et al, Eur J Cancer, 2017)
* Age ≥18 years
* Have failed at least one previous line of systemic therapy
* Have received mogamulizumab in real life setting after the approval and reimbursement of the drug from the National Health System in December 2020
* Have received first dose of mogamulizumab between 01/01/2021 and 31/01/2023
* Have received mogamulizumab at the standard approved dose (1.0 mg/kg intravenously on days 1, 8, 15 and 22 of the first cycle and on days 1 and 15 of subsequent cycles)
* Availability of complete medical records.

Exclusion Criteria:

• Patients not meeting the above-mentioned inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by relapsed/refractory Cutaneous T-cell Lymphoma who have received Mogamulizumab in real life settings
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
To assess Overall response rate lasting at least 4 months (ORR4) | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Overall response lasting at least 4 months from response (CR+PR) to treatment with mogamulizumab

SECONDARY OUTCOMES:
To assess Frequencies of baseline characteristic compared with the expected from MAVORIC study | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  To identify whether real life patients show baseline characteristics (i.e., CTCL subtype, cutaneous and blood involvement, staging) in line with the population enrolled in the MAVORIC trial
To assess Overall response rate (ORR) at 1 month, ORR at 4 months and best ORR obtained from beginning of treatment with Mogamulizumab | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  Evaluate the early and late activity of mogamulizumab
To assess Logistic regression of ORR4 with peripheral blood involvement score | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  To identify whether the presence of a B1 B2 score is associated with a higher response rate in the skin, compared to B0
To assess Frequencies of adverse events collected with the clinical course | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  To investigate whether the presence of a cutaneous side effect is associated with a different clinical course and high response rate
To assess Progression Free Survival (PFS), Overall Survival (OS), Time to Next Treatment (TTNT) | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  To investigate the overall efficacy of treatment. Time to event functions will be stratified according to the disease subtype (Mycosis fungoides/Sézary syndrome), stage (early vs advanced), number of previous treatment lines (1 or more than)
To assess Frequencies of patients who receive mogamulizumab as bridge to allotransplant, as well as disease features of these patients and type of response to transplant | The endpoint will be evaluated from the beginning to the end of the study (up to 18 months)
  To evaluate the number and related disease features of patients who receive mogamulizumab as bridge to allotransplant, as well as the type of response to transplant in these patients

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Quaglino, MD, Principal Investigator — SC Dermatologia U - A.O.U. Città della Salute e della Scienza di Torino
Locations (21):
- Italy (21):
  - Clinica di Ematologia - AOU Ospedali Riuniti delle Marche, Ancona
  - S.C. Ematologia e Trapianto emopoietico - A.O. S.Giuseppe Moscati, Avellino
  - Clinica Dermatologia - A.O.U. Policlinico Consorziale, Bari
  - U.O.C. Ematologia - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Istituto di Ematologia - Policlinico S.Orsola-Malpighi, Bologna
  - S.C. Ematologia - ASST Spedali Civili, Brescia
  - S.C. Ematologia e CTMO - A.O. Brotzu Ospedale Businco, Cagliari
  - U.O.C. di Ematologia - A.O.U. Policlinico S. Marco, Catania
  - Unità funzionale di Ematologia - Azienda Ospedaliera Universitaria Careggi, Florence
  - S.C. Dermatologia - IRCCS Policlinico S. Martino, Genova
  - S.C. Ematologia e Terapie Cellulari - IRCCS Policlinico S. Martino, Genova
  - U.O.C. Dermatologia - Ospedale Maggiore Policlinico Fondazione IRCCS Ca' Granda, Milan
  - Clinica Dermatologica - A.O.U. Luigi Vanvitelli, Napoli
  - U.O.C. Dermatologia . A.O.U. di Padova, Padua
  - Divisione di Ematologia - IRCCS Policlinico San Matteo, Pavia
  - U.O. Ematologia - Ospedale Guglielmo da Saliceto, Piacenza
  - U.O.C. Ematologia - Policlinico Tor Vergata, Roma
  - UOSD Porfirie e Malattie Rare - IRCCS I.F.O. San Gallicano, Roma
  - U.O.C. Ematologia - A.O.U. Senese, Siena
  - S.C. Dermatologia U - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - Verona - AOU Integrata di Verona - U.O. Ematologia, Verona